CLINICAL TRIAL: NCT00647491
Title: A Study of Adalimumab in Adult Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M02-575
Record Dates: First submitted 2008-03-27; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 20 mg (Experimental): 20 mg adalimumab eow
  Interventions: Biological: adalimumab
- 40 mg (Experimental): 40 mg adalimumab eow
  Interventions: Biological: adalimumab
- 80 mg (Experimental): 80 mg adalimumab eow
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator): Placebo eow
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab — 20 mg sc eow
  Other Names: ABT-D2E7; Humira
  Arms: 20 mg
Biological: adalimumab — 40 mg sc eow
  Other Names: ABT-D2E7; Humira
  Arms: 40 mg
Biological: adalimumab — 80 mg sc eow
  Other Names: ABT-D2E7; Humira
  Arms: 80 mg
Biological: placebo — placebo sc eow
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety, efficacy and pharmacokinetics of three doses of adalimumab in adult Japanese subjects with RA

ELIGIBILITY:
Inclusion Criteria:

* Meet ACR criteria for diagnosis of active RA and have at both screening and baseline visits >10 swollen joints, >12 tender joints.
* Subjects must have failed prior treatment with one or more DMARDs.
* A negative (serum) pregnancy test for all female subjects of child-bearing potential at screening and a negative (urine) pregnancy test prior to study drug administration.
* Body weight less than or equal to 100 kg

Exclusion Criteria:

* A history of, or current, acute inflammatory joint disease of different origin from RA.
* Prior treatment with any TNF antagonist, including adalimumab.
* Any ongoing chronic or active infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics.
* Unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke or any poorly controlled medical condition.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2004-02; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
ACR20 | Week 24

SECONDARY OUTCOMES:
ACR20 | Week12
ACR50 | Weeks 12 and 24
ACR70 | Weeks 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, Ph.D., Study Director — Abbott
Locations (25):
- Japan (25):
  - Aichi
  - Chiba
  - Ehime
  - Fukui
  - Fukuoka
  - Gunma
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Ishikawa
  - Kagoshima
  - Kanagawa
  - Kyoto
  - Miyagi
  - Nagano
  - Nagasaki
  - Niigata
  - Okayama
  - Osaka
  - Saitama
  - Shizuoka
  - Tochigi
  - Tokushima
  - Tokyo
  - Toyama

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778